CLINICAL TRIAL: NCT03852667
Title: The Effect of Secondary Prevention for Low Back Pain by Means of Pain Education and Exercise Therapy in Patients With Recurrent Low Back Pain
Brief Title: The Effect of Secondary Prevention in Patients With Recurrent Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EC/GK2017/1508
Record Dates: First submitted 2019-01-24; First posted 2019-02-25 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Low Back Pain, Recurrent
Keywords: low back pain; recurrent; non-specific; secondary prevention; pain neuroscience education; exercise therapy
MeSH Terms: conditions — Low Back Pain; Recurrence | interventions — Exercise Therapy

STUDY DESIGN:
Intervention Model Description: The randomization schedule was extracted from the website www.sealedenvelope.com . The randomization was expected to have the same amount of one gender in each group. The control group was group A, the group that only received PNE was group B and the group who received PNE and exercise therapy was group C.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The leading investigators, as well as the outcome assessors are masked and do not know to which arm the subjects are allocated to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): No intervention between the two test sessions
- Pain Neuroscience Education (Active Comparator): Two sessions (30 min) of Pain Neuroscience Education
  Interventions: Behavioral: Pain Neuroscience Education
- Pain neuroscience education - exercise (Experimental): 2 sessions of PNE and 5 sessions of exercise therapy.
  Interventions: Behavioral: Pain Neuroscience Education; Other: Exercise therapy

INTERVENTIONS:
Behavioral: Pain Neuroscience Education — The PNE intervention consisted of 2 sessions of 30 minutes. In the first session, the main goal is to explain the patient why pain is important and why people can't live without it. Besides it is explained why objective findings such as x-rays, MRI, CT scans, etc. often lack significant findings despite the pain that the patient experiences. This first session of pain education might help the patient understand that pain is necessarily a result from tissue damage. Furthermore, the session explains the right approach to conquer pain and to avoid going down in this vicious circle of low back pain. The second session of PNE, is a revision of the first session, continuing on what was unclear from the first session.
  Arms: Pain Neuroscience Education; Pain neuroscience education - exercise
Other: Exercise therapy — The exercise therapy varies form analytical exercises in the first sessions, to functional and sports related exercises near the following sessions. The first session focuses on the lumbar neuromuscular control of the patients: first a voluntary contraction of the Transversus Abdominis muscle, the Multifidus muscle and the pelvic floor muscles is learned. When the subject is able to maintain the combined contraction for 10 times, the exercises evolve to more complicated tasks. In the final stage, more functional and sport specific tasks will be exercised.
  Arms: Pain neuroscience education - exercise

SUMMARY:
This study investigates the effect of a secondary intervention program for low back pain in patients with recurrent low back pain. One third of the subject will receive no therapy, one third wil receive 2 sessions of pain neuroscience education (PNE) and one third will receive two sessions of PNE and 5 sessions of exercise therapy over 6 weeks.

DETAILED DESCRIPTION:
Participants:

60 individuals with recurrent non-specific LBP were recruited through advertisement in sport facilities, social media and among friends and family.

Testing:

The testing was performed before and after a six week period by three blinded 2nd master students of physiotherapy of University of Ghent. The pre and post testing were almost identical and lasted 1 hour, only for the first testing an anamnesis was conducted to evaluate inclusion and exclusion criteria. The identical parts were tests for motor control, muscle performance and psychosocial factors.

Intervention:

The subjects were divided into 3 groups, only group B and C were given treatment. Group B had 2 sessions PNE over a period of two weeks. Group C received 2 sessions of PNE and 5 sessions of exercise therapy over a period of six weeks. Each of the sessions lasted 30 minutes and took place at the clinical practice room at the university of Ghent. Group C began the exercise therapy a week after the second session of PNE.

ELIGIBILITY:
Inclusion Criteria:

* In remission during testing
* recurrent low back pain (RLBP) >6months
* 2 or more episodes in the past year
* Pain flare of ≥24 hours, characterized by an increase of ≥2 on an Numeric Rating Scale (NRS) scale and/or ≥5 on the Roland Morris Disability Questionnaire
* Followed by a pain-free episode of ≥1 month, characterized by a 0/10 on an NRS scale and/or <2 on the Roland Morris Disability Questionnaire
* Non-specific RLBP (no cause for Low back pain (LBP); >3y post discus herniation)
* 1 year or more post-natal

Exclusion Criteria:

* Use of antidepressants or analgesics (except for NSAIDs or paracetamol), taken 2 weeks before the testing
* Neurologic, respiratory, circulatory, or severe orthopedic diseases
* Pregnancy
* Specific LBP causes
* A history of cognitive exercise therapy and/or specific motor control training
* current treatment or new therapies starting <6 weeks before baseline assessment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2019-09-29 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Quality of core movement control by use of the Luomajoki test battery | 6 weeks
  A core movement control test battery is performed pre and post intervention, to assess a possible movement control dysfunction of the low back. This test battery consists out of six tests: waiters bow, dorsal tilt of pelvis actively in upright standing, one leg stance, sitting knee extension test, quadruped position, prone lying active knee flexion.
Quality of proprioception of the core by use of the lumbopelvic position-reposition test | 6 weeks
  A lumbopelvic position-reposition test was performed pre and post intervention for measuring proprioceptive deficits in the core in the subjects. This repositioning test evaluates the participant's repositioning accuracy of the pelvis, low back and trunk after a dynamic task.
Quality of neuromuscular control by use of the lumbopelvic movement control test | 6 weeks
  The neuromuscular control of the lumbar region is measured pre and post intervention. This test evaluates a repeated lumbopelvic movement on five categories; quality of the lumbopelvic motion, control of the adjacent areas, preference of motion direction, breathing, and the amount of good quality repetitions.

SECONDARY OUTCOMES:
Improvement of trunk strength by use of a hand held dynamometer | 6 weeks
  The maximal voluntary contraction of the extensor and flexor muscles of the back will be assessed pre and post intervention, using a hand-held dynamometer. This measurement will provide an insight on the total muscle strength.
Psychosocial factor "Tampa scale of kinesiophobia" | 6 weeks
  The clinical questionnaire "Tampa scale of kinesiophobia" was used to assess the the amount of pain related anxiety in low back pain, pre and post intervention. This scale contains 17 items rated on a 4-point Likert scale (ranging from 1= highly agree to 4 highly disagree). A higher total score means a higher amount of fear of movement.
Psychosocial factor "Pain catastrophizing scale" | 6 weeks
  The clinical questionnaire "Pain catastrophizing scale" was used to assess the amount of catastrophizing pre and post intervention. The PCS contains 13 items rated on a 5-point Likert scale (ranging from 0 =not at all to 4 =all the time). The total score and 3 subscale scores are measured (rumination, magnification and helplessness) with subscale scores ranging between 0-16, 0-12, and 0-24, respectively. A score ≥11 for rumination, ≥5 for magnification, ≥13 for helplessness or a total score of ≥30 are clinically relevant cut offs for identifying pain catastrophizing.
Psychosocial factor "Pain disability index" | 6 weeks
  The clinical questionnaire "pain disability index" was used to assess the degree of interruption of activities from daily life due to pain in the previous week, pre and post intervention. The PDI contains 7 items scored on a Likert scale with scores ranging between 0 (=no disability at all) and 10 (=affectation or disruption of an individual's ability to participate in activities due to pain). Higher scores indicate more pain related disability.
Psychosocial factor "Multidimensional pain inventory" | 6 weeks
  The clinical questionnaire "Multidimensional pain inventory" was used to assess the different aspects of pain and their influence on daily life experiences pre and post intervention. The MPI contains 28 items rated on a 7-point Likert scale (ranging from 0 to 6). All 28 items are divided among 5 subscales (pain severity, perceived life control and affective distress, interference with the daily life due to present pain complaint and social support). A higher score on the social support and life control subscales represents a better outcome. A higher score on the subscales interference in daily life, pain severity and affective distress represents a less favourable outcome.
Psychosocial factor "Roland Morris disability questionnaire" | 6 weeks
  The clinical questionnaire was used to assess the disability due to low back pain in the last 24 hours, pre and post intervention. The RMDS contains 24 statements. The patient is instructed to put a mark next to each appropriate statement and all marks are added up. Greater levels of disability are reflected by higher numbers on a 24-point scale. A difference of ≥5 indicates a clinical important change.

CONTACTS AND LOCATIONS:
Overall Officials: Lieven Danneels, PhD, Study Chair — University Ghet
Locations (1):
- Vakgroep Revalidatiewetenschappen, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: No